CLINICAL TRIAL: NCT05688332
Title: Comparison of Glycaemic and Cardiovascular Treatment Outcomes of Voglibose Versus Glibenclamide Added to Metformin in T2DM Patients in Zambia: An Open-label Randomised Clinical Trial
Brief Title: Glycaemic & Cardiovascular Treatment Outcomes of Voglibose Vs Glibenclamide Added to Metformin in T2DM Patients
Acronym: VMGMProtocol
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Zambia (Other)
Collaborators: University Teaching Hospital, Lusaka, Zambia (Other)
Responsible Party: Principal Investigator, Lawrence Mukela, Principal Investigator, University of Zambia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202112030076; IRB Number: 00011000 (Other: UNZAHSREC); IORG Number: 0009227 (Other: UNZAHSREC); FWA Number: 00026270 (Other: UNZAHSREC)
Record Dates: First submitted 2022-12-27; First posted 2023-01-18 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Diabetes Mellitus Type 2 Without Complication
Keywords: voglibose; Metformin; Glibenclamide; Outcomes
MeSH Terms: interventions — voglibose; Metformin; Glyburide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Voglibose + Metformin (Group B) (Experimental): In the B treatment group, 59 participants will be randomly assigned to initially voglibose 0.2mg TDS immediately before meals + metformin 500mg BD immediately before meals daily. Individual drug doses will be adjusted to the next higher doses after 6 to 12 days, at next clinical visits based on home based recorded blood glucose profiles. The maximum daily recommended dose of metformin of 2g and voglibose 0.9mg will not be exceeded.
  Interventions: Drug: Voglibose + Metformin
- Glibenclamide + Metformin (Group A) (Active Comparator): In treatment group A, 59 participants will initially be randomly allocated by study team members to the glibenclamide 5mg O.D + metformin 500mg BD regimen.
  In this study, 10mg glibenclamide and 2g metformin will not be exceeded daily.
  Interventions: Drug: Glibenclamide + Metformin

INTERVENTIONS:
Drug: Voglibose + Metformin — In treatment group B, 59 participants will also be randomly assigned to the voglibose 0.2/0.3mg TDS + metformin 500mg BD treatment combination to be taken orally daily, during or immediately after meals with dose titration at day 6 and 12 if the average fasting blood glucose (FBG) level is ≥7 mmol/L (126 mg/dL) and then dosage will be maintained for the remainder of the treatment period Participants in the intervention group initially receiving voglibose 0.2mg + metformin 500mg BD will be dose-titrated to voglibose 0.3mg +metformin 1g BD.
  The duration of therapy for each participant will be 12 weeks, which is the minimum period for evaluating the primary endpoint.
  Arms: Voglibose + Metformin (Group B)
Drug: Glibenclamide + Metformin — The drugs (glibenclamide + metformin), in the control or comparator group will also be taken orally, glibenclamide once a day (OD) before meals, and metformin twice a day (BD) also before meals. These drugs will also be taken with a dose-titration at days 6 and 12 if the average is FBG level will be ≥ 7 mmol/L and the dose will be maintained for the remainder of the study period.
  The duration of therapy for each participant will be 12 weeks, which is the minimum period for evaluating the primary endpoint. In this group, participants will initially receive glibenclamide 5mg once daily (OD) + metformin 500mg BD then will be dose-titrated to glibenclamide 10mg OD + metformin 1g BD.
  Arms: Glibenclamide + Metformin (Group A)

SUMMARY:
The goal of this clinical trial is to compare blood-sugar control and blood circulatory system risk-position in type 2 diabetes patients on voglibose versus those on glybenclamide when the two drugs are added to metformin because metformin alone is not controlling the blood-sugar well. The results of this trial will help in improving the health and treatment results of the type 2 diabetic patients.

The main question the trial aims to answer is whether there is a difference in blood-sugar and blood circulatory system treatment results between voglibose + metformin and glibenclamide + metformin treatment combinations.

Participants that agree to participate in the trial will be asked to provide a sample of blood so that the following measurable laboratory factors will be used to compare any differences in treatment results between the two treatment groups from the beginning to the end of the trial:

* Total Cholesterol (TC),
* Low Density Lipoproteins (LDL-c),
* High Density Lipoproteins (HDL-c),
* Fasting Triglycerides (FTG),
* Fasting blood sugar (FBS),
* Post prandial blood sugar (PPBG),
* Glycated hemoglobin (HbA1c) correlated to hemoglobin level,
* creatinine,
* blood urea and
* electrolytes (K+, Na+, Cl-).

DETAILED DESCRIPTION:
BACKGROUND: Diabetes is an increasingly important risk factor for CVD. Individuals with it continually have an increased risk of CV caused mortality. It can be classified as T1DM, T2DM, GDM and others. Metformin is a T2DM 1st line Oral Hypoglycaemic Agent (OHA). It usually requires a 2nd line add-on drug if blood glucose control is not on target. The add-on drug can either be insulin, an injectable incretin mimetic, or an OHA. The choice of the OHA should be considered with regard to improving the glycaemic control as well as reducing the CVD risk. Glibenclamide, a Sulphonylurea (SU), is a commonly used OHA in Zambia. It is associated with hypoglycaemia and arrhythmias. On the other hand voglibose, an alpha glucosidase inhibitor (AGI), is not associated with hypoglycaemia or with negative CV events. AGIs are associated with reduced PPBG by reducing the absorption of glucose in the GI tract after a carbohydrate meal. Reduced PPBG prevents macrovascular complications. Since maize (a carbohydrate) is a staple food in Zambia, there is need to investigate the glycaemic control in patients with T2DM using voglibose which is as affordable as glibenclamide.

MAIN AIM: To investigate the extent of glycaemic control and CV risk parameter effects of voglibose versus glibenclamide add-on therapies in Zambian patients with T2DM as we do not have published studies on these parameters in our patients.

METHOD: This study will be a 12 weeks dual-center open-label randomised clinical trial to comparatively evaluate the glycaemic and CV treatment outcomes of voglibose vs glibenclamide add-on therapies in native Zambian patients with T2DM inadequately controlled on 1g/day of metformin monotherapy. In this study, glycaemic and CV parameters will be quantified and classified in the laboratory to determine extent of glycaemic control and CVD risk reduction. Participants to be included will be male and female native Zambian patients aged 22 to 59 years on metformin monotherapy for at least 12 weeks with HbA1c > 7.0%. They will be randomly allocated by study team members to two treatment arms i.e., the voglibose-metformin or the glibenclamide-metformin regimen in a 1:1 computer generated simple randomisation. The participants will then be followed up to the 6th and 12th week for data collection prior to comparative analysis of the expected outcome.

EXPECTED OUTCOME: Change in glycaemic and CV parameters in the two groups after 6 and 12 weeks of add-on therapy.

SIGNIFICANCE: To help determine the glycaemic and CV risk status of patients with T2DM on voglibose and glibenclamide, thereby ascertain improvement in their healthcare and treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* In order to be eligible to participate in this study, an individual must meet all of the following criteria:

  * Provision of signed and dated informed consent form.
  * Stated willingness to comply with all study1 procedures and availability for the durtion of the study.
  * Male or female, aged 22-59 years.
  * In good general health as evidenced by medical history, diagnosed with T2DM and on tolerated dose of at least 2g/day of metformin monotherapy.
  * Ability to take oral medication and be willing to adhere to the medication regimen through out the study period.
  * For females of reproductive potential use of highly effective contraception.
  * Native-Zambian participants
  * Must be on metformin monotherapy for 12 weeks or longer.
  * Glycated haemoglobin (HbA1c) must be >7.0% within 12 weeks before screening.

Exclusion Criteria:

* An individual who meets any of the following criteria will be excluded from participation in this study:

  * Hypersensitivity or contraindication to AGIs
  * Hypersensitivity or contraindication to SUs
  * Type 2 diabetes patients with pregnancy or lactation
  * Patients with acute complications like diabetic ketoacidosis, or hyperosmolar hyperglycaemic state at the time of screening
  * Patients with established cardiovascular disease, e.g.; HF, coronary artery disease
  * Patients with altered haemoglobin levels, e.g.; in conditions like anaemias and haemoglobimopathies such as thalassemia
  * Patients on concomitant corticosteroid therapy.

Ages: 22 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 118 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
Change in mean Glycated Hemoglobin (HbA1c) levels | Baseline & Week 6
  The null hypothesis is that there is no significant difference between the voglibose and glibenclamide treatment groups in the change in mean HbA1c levels after 6 weeks of add-on therapy to metformin in the T2DM patients (i.e. H0: µ1 = µ2 where µ1 is the mean HbA1c change in the glibenclamide group and µ2 is the mean HbA1c change in the voglibose group). The alternative hypothesis is that there is a significant difference between the voglibose and glibenclamide groups in the change in mean HbA1c levels after 6 weeks of add-on therapy to metformin in the T2DM patients (i.e. H1: µ1 ≠ µ2).
Change in mean Glycated Hemoglobin (HbA1c) levels | Baseline & Week 12
  The null hypothesis is that there is no significant difference between the voglibose and glibenclamide treatment groups in the change in mean HbA1c levels after 12 weeks of add-on therapy to metformin in the T2DM patients (i.e. H0: µ1 = µ2 where µ1 is the mean HbA1c change in the glibenclamide group and µ2 is the mean HbA1c change in the voglibose group). The alternative hypothesis is that there is a significant difference between the voglibose and glibenclamide groups in the change in mean HbA1c levels after 12 weeks of add-on therapy to metformin in the T2DM patients (i.e. H1: µ1 ≠ µ2).

SECONDARY OUTCOMES:
Change in Glycemic control with regard to Fasting Plasma Glucose (FPG) | Baseline & week 6
  Differences in change in glycemic control with regard to FPG: The null hypothesis is that there is no significant difference between the voglibose and glibenclamide treatment groups in the mean FPG change (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean FPG change in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between the voglibose and glibenclamide groups in the mean changes of FPG (i.e. H1: µ1 ≠ µ2).
Change in glycemic control with regard to Fasting Plasma Glucose (FPG) | Baseline & week 12
  Differences in change in glycemic control with regard to FPG: The null hypothesis is that there is no significant difference between the voglibose and glibenclamide treatment groups in the mean FPG change (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean FPG change in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between the voglibose and glibenclamide groups in the mean changes of FPG (i.e. H1: µ1 ≠ µ2).
Change in glycemic control with regard to Post Prandial Blood Glucose (PPBG) | Baseline & week 6
  Differences in Change in glycemic control with regard to PPBG: The null hypothesis is that there is no significant difference between the voglibose and glibenclamide treatment groups in the mean PPBG change (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean PPBG change in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between the voglibose and glibenclamide groups in the mean changes of PPBG (i.e. H1: µ1 ≠ µ2).
Change in glycemic control with regard to Post Prandial Blood Glucose (PPBG) | Baseline & week 12
  Differences in change in glycemic control with regard to PPBG: The null hypothesis is that there is no significant difference between the voglibose and glibenclamide treatment groups in the mean PPBG change (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean PPBG change in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between the voglibose and glibenclamide groups in the mean changes of PPBG (i.e. H1: µ1 ≠ µ2).
Lipid profile (LDL-c, HDL-c, TC, TG) comparison | Baseline & Week 6
  Lipid profile (LDL-c, HDL-c, TC, TG) comparison: The null hypothesis is that there is no difference between the voglibose and glibenclamide groups in the mean changes in lipid profile (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean changes in lipid profile in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between voglibose and glibenclamide groups in the mean changes in lipid profile (i.e. H1: µ1 ≠ µ2).
Lipid profile (LDL-c, HDL-c, TC, TG) comparison | Baseline & Week 12
  Lipid profile (LDL-c, HDL-c, TC, TG) comparison: The null hypothesis is that there is no difference between the voglibose and glibenclamide groups in the mean changes in lipid profile (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean changes in lipid profile in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between voglibose and glibenclamide groups in the mean changes in lipid profile (i.e. H1: µ1 ≠ µ2).
Anthropometric parameter changes in BMI | Baseline & Week 6
  Anthropometric parameter changes in BMI: The null hypothesis is that there is no difference between the voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean anthropometric parameter changes in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H1: µ1 ≠ µ2).
Anthropometric parameter changes in BMI | Baseline & Week 12
  Anthropometric parameter changes in BMI: The null hypothesis is that there is no difference between the voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean anthropometric parameter changes in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H1: µ1 ≠ µ2).
Anthropometric parameter changes in Waist Circumference (WC) | Baseline & Week 6
  Anthropometric parameter changes in WC: The null hypothesis is that there is no difference between the voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean anthropometric parameter changes in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H1: µ1 ≠ µ2).
Anthropometric parameter changes in Waist Circumference (WC) | Baseline & Week 12
  Anthropometric parameter changes in WC: The null hypothesis is that there is no difference between the voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H0: µ1 = µ2 where µ1 and µ2 represent the mean anthropometric parameter changes in the glibenclamide and voglibose groups respectively). The alternative hypothesis is that there is a difference between voglibose and glibenclamide groups in the mean anthropometric parameter changes (i.e. H1: µ1 ≠ µ2).
Drug related AEs | Baseline & Week 6
  Drug related AEs: The null hypothesis is that there is no difference between the proportion of participants experiencing drug related AEs in the voglibose and glibenclamide groups (i.e. H0: p1 = p2 where p1 and p2 represent the proportion of participants experiencing a drug related AE in the glibenclamide and voglibose groups, respectively). The alternative hypothesis is that there is a difference between the proportion of participants experiencing drug related AEs in the voglibose and glibenclamide groups (i.e. H1: p1 ≠ p2).
Drug related AEs | Baseline & Week 12
  Drug related AEs: The null hypothesis is that there is no difference between the proportion of participants experiencing drug related AEs in the voglibose and glibenclamide groups (i.e. H0: p1 = p2 where p1 and p2 represent the proportion of participants experiencing a drug related AE in the glibenclamide and voglibose groups, respectively). The alternative hypothesis is that there is a difference between the proportion of participants experiencing drug related AEs in the voglibose and glibenclamide groups (i.e. H1: p1 ≠ p2).

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in diabetes mellitus. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting parties.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact lawrencemukela@gmail.com

REFERENCES:
- [Background] American Diabetes Association Professional Practice Committee. 2. Classification and Diagnosis of Diabetes: Standards of Medical Care in Diabetes-2022. Diabetes Care. 2022 Jan 1;45(Suppl 1):S17-S38. doi: 10.2337/dc22-S002. PMID 34964875
- [Background] Rosenquist KJ, Fox CS. Mortality Trends in Type 2 Diabetes. In: Cowie CC, Casagrande SS, Menke A, Cissell MA, Eberhardt MS, Meigs JB, Gregg EW, Knowler WC, Barrett-Connor E, Becker DJ, Brancati FL, Boyko EJ, Herman WH, Howard BV, Narayan KMV, Rewers M, Fradkin JE, editors. Diabetes in America. 3rd edition. Bethesda (MD): National Institute of Diabetes and Digestive and Kidney Diseases (US); 2018 Aug. CHAPTER 36. Available from http://www.ncbi.nlm.nih.gov/books/NBK568010/ PMID 33651566
- [Background] Coleman RL, Scott CAB, Lang Z, Bethel MA, Tuomilehto J, Holman RR. Meta-analysis of the impact of alpha-glucosidase inhibitors on incident diabetes and cardiovascular outcomes. Cardiovasc Diabetol. 2019 Oct 17;18(1):135. doi: 10.1186/s12933-019-0933-y. PMID 31623625
- [Background] Akmal M, Patel P, Wadhwa R. Alpha Glucosidase Inhibitors. 2024 Feb 28. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2025 Jan-. Available from http://www.ncbi.nlm.nih.gov/books/NBK557848/ PMID 32496728